CLINICAL TRIAL: NCT07120776
Title: Positron Emission Tomography to Assess the Effect of Camzyos on Ischaemia in Hypertrophic Obstructive Cardiomyopathy: The PEACH Trial
Brief Title: Positron Emission Tomography to Assess the Effect of Camzyos on Ischaemia in HOCM: PEACH Trial
Acronym: PEACH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Andrew Crean, Professor, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS Project ID: 349544; REC Reference 25/ES/0044 (Other: East of Scotland Research Ethics Service (EoSRES))
Record Dates: First submitted 2025-08-01; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy (HOCM); Left Ventricular Outflow Tract Obstruction; Myocardial Ischaemia
Keywords: Camzyos; Mavacamten; HOCM; HCM; Cardiac PET; Rubidium-82 PET-CT; Myocardial Perfusion; Nuclear cardiology; Left ventricular outflow obstruction; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Ventricular Outflow Obstruction, Left; Coronary Artery Disease; Cardiomyopathies | interventions — MYK-461

STUDY DESIGN:
Intervention Model Description: Single-arm prospective cohort study of patients with HOCM undergoing PET imaging before and after Camzyos treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Camzyos (Mavacamten) Treatment Group (Experimental): Patients with Hypertrophic Obstructive Cardiomyopathy (HOCM) who are clinically prescribed Camzyos (Mavacamten) as part of standard care. Participants will undergo baseline(standard care) and 12-month follow-up (research scan) myocardial perfusion PET-CT scans to assess the effect of Camzyos on myocardial ischaemia.
  Interventions: Drug: Camzyos (Mavacamten)

INTERVENTIONS:
Drug: Camzyos (Mavacamten) — Camzyos (Mavacamten), a selective cardiac myosin inhibitor prescribed as part of routine care in patients with symptomatic HOCM. The study evaluates its effect on myocardial perfusion over a 12-month period using PET-CT imaging.

SUMMARY:
Hypertrophic obstructive cardiomyopathy (HOCM) is a heritable heart condition that leads to the thickening of the heart muscle and causes obstruction of blood flow, impeding it's ejection from the heart (LVOT obstruction). Often individuals with HOCM suffer from chest pain and shortness of breath due to lack of oxygen supply (ischaemia) to the heart muscle in the absence of blockages in the coronary arteries.

Despite proven advances in treatment of LVOT obstruction with the novel medication Camzyos (Mavacamten), there is a limited understanding of its effect on myocardial ischaemia.

This study, called the PEACH Trial, is designed to assess whether Camzyos also improves blood supply (perfusion) to the heart muscle in patients with HOCM. A specialised imaging technique called Positron Emission Tomography/Computed Tomography (PET-CT), using Rubidium-82 will be used to evaluate blood flow to the heart muscle before and after treatment. Camzyos is part of participants' regular clinical treatment and is not being supplied, administered, or influenced by the study in any way.

Participants with HOCM who are starting treatment with Camzyos as part of their clinical care will undergo a baseline PET-CT scan (if not already done), and a second scan after 12 months. The follow-up scan is done solely for research purposes. The scans will allow researchers to evaluate whether the medication improves myocardial perfusion in addition to relieving outflow obstruction.

The study is sponsored by the University of Manchester and funded by Bristol Myers Squibb. It will involve up to 75 participants recruited at Manchester University NHS Foundation Trust. The findings could help improve understanding of how Camzyos works and support personalised treatment approaches in HOCM.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Aged 18 and over.
3. Confirmed diagnosis of Hypertrophic Obstructive Cardiomyopathy (HOCM) based on diagnostic criteria, such as unexplained left ventricular hypertrophy with a maximal wall thickness ≥15 mm in the absence of uncontrolled hypertension, valvular heart disease, or HCM phenocopies such as amyloidosis and storage disorders, and presence of either a resting or provoked peak left ventricular outflow tract (LVOT) gradient ≥30 mmHg.
4. Symptoms suggestive of myocardial ischaemia (chest pain, shortness of breath on exertion) with a clinical indication for Rb-PET.
5. Eligible for Mavacamten treatment according to standard clinical guidelines. [see: https://www.nice.org.uk/guidance/ta913/chapter/1-Recommendations]. Mavacamten is part of participants' regular clinical treatment and is not being supplied, administered, or influenced by the study in any way.
6. PET-CT performed for clinical reasons at any time in the preceding 18 months if reported as abnormal.

Exclusion Criteria:

1. Patients with obstructive coronary artery disease (epicardial coronary stenosis >50%, assessed by either invasive coronary angiography or computed tomography angiography (CTCA). Patients will undergo the initial PET study as part of their routine clinical care. If evidence of ischaemia is identified, the standard next step would involve either CT coronary angiography or, in some cases, invasive angiography to guide further clinical management. If the angiography reveals a clear lesion responsible for the ischaemia identified on PET, the patient will not be eligible for inclusion in the study and will not be approached. Conversely, if the angiography does not identify a definitive cause for the ischaemia, it will be presumed to be of microvascular origin. In such cases, the patient becomes eligible for the study and will be approached to discuss participation and provide consent at this stage. It is important to emphasize that any angiographic procedure occurs prior to consent and as part of routine clinical care. No angiographic investigations are planned or conducted as part of the study protocol. Data from the clinical angiogram will not be included in the study, except to note a 'positive angiogram' as a reason for patient exclusion.
2. Contraindications to Mavacamten, including left ventricular ejection fraction (LVEF) less than 55%, hypersensitivity or allergic reaction to the drug.
3. Contraindication to Rubidium PET-CT, including:

   * Pregnancy or breastfeeding.
   * Severe claustrophobia.
   * Morbid obesity when the patient dimensions are beyond the scanning chamber capacity.
4. Any medical condition, which in the opinion of the Investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in Myocardial Ischaemia: | 12 months
  This will be assessed using Rubidium PET-CT. Looking at change in parameters such as global myocardial blood flow reserve (GMBFR)
Change in Myocardial Ischaemia: | 12 months
  This will be assessed using Rubidium PET-CT. Looking at change in parameters such as global myocardial stress flow (GMSF).
Change in Myocardial Ischaemia: | 12 months
  This will be assessed using Rubidium PET-CT. Looking at change in parameters such as coronary flow capacity (CFC).

SECONDARY OUTCOMES:
Patient-Reported Symptoms | 12 months
  Secondary outcomes:
  1. Patient-Reported Symptoms:
  • Angina and Shortness of Breath: Changes in the frequency and severity of angina episodes and shortness of breath will be documented using validated the Seattle Angina Questionnaire- 7 (SAQ).
  Seattle Angina Questionnaire-7 (SAQ-7, 2014 version):
  The SAQ-7 is a validated, patient-reported outcome measure assessing the impact of angina on health status. It consists of 7 items covering 3 domains: Physical Limitation, Angina Frequency, and Quality of Life. Each domain is scored on a 0-100 scale, where higher scores indicate better health status (less angina, fewer physical limitations, and improved quality of life). Scores are transformed according to published scoring algorithms. The SAQ-7 Summary Score is the mean of the 3 domain scores.
  Minimum score: 0 (worst possible angina-related health status) Maximum score: 100 (no angina, no limitation, best possible quality of life)
Patient-Reported Symptoms | 12 months
  Secondary outcomes:
  1. Patient-Reported Symptoms:
  * Angina and Shortness of Breath: Changes in the frequency and severity of angina episodes and shortness of breath will be documented using validated the the HCM Shortness of Breath Questionnaire (HCMSQ-SoB) (also used in the EXPLORER-HCM trial)
  * The HCMSQ total score is as the equally weighted sum of the three domain scores, i.e., the sum of the SoB domain score divided by four (items), the tiredness domain score (a single item), and the CV symptom domain score divided by three (items), if all three domain scores are calculated; otherwise, the HCMSQ total score is missing. The potential range of scores is 0-12.5, with lower scores indicating a lower presence of symptoms overall/better health.
Patient-Reported Symptoms | 12 months
  Secondary outcomes:
  NYHA Functional Class: Improvement in NYHA functional class will be evaluated to assess changes in functional capacity and symptom severity.
  New York Heart Association (NYHA) Functional Classification - Ordinal scale ranging from Class I (no symptoms and no limitation in ordinary physical activity) to Class IV (severe limitations; symptoms present even at rest). Lower classes indicate better functional status, and improvement is reflected by a decrease in NYHA class from baseline.
Subgroup Analyses | 12 months
  Differences in Efficacy Based on Patient Subgroups:
  • Subgroup Analyses: The study will investigate differences in the impact of Mavacamten on myocardial ischemia and symptoms based on:
  o Age years (younger vs. older patients)
Subgroup Analyses | 12 months
  Differences in Efficacy Based on Patient Subgroups:
  • Subgroup Analyses: The study will investigate differences in the impact of Mavacamten on myocardial ischemia and symptoms based on:
  o Sex (male vs. female)
Subgroup Analyses | 12 months
  Differences in Efficacy Based on Patient Subgroups:
  • Subgroup Analyses: The study will investigate differences in the impact of Mavacamten on myocardial ischemia and symptoms based on:
  o Genetic Status (gene-positive vs. gene-negative vs VUS)
Subgroup Analyses | 12 months
  Differences in Efficacy Based on Patient Subgroups:
  • Subgroup Analyses: The study will investigate differences in the impact of Mavacamten on myocardial ischemia and symptoms based on:
  o Baseline LVOT Gradient Levels (mmHg) (higher vs. lower LVOT gradients)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Crean, BSc BM MRCP FRCR MPhil MPH, Principal Investigator — University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data access is limited to the research team as per ethical and institutional approvals.

REFERENCES:
- [Background] Olivotto I, Oreziak A, Barriales-Villa R, Abraham TP, Masri A, Garcia-Pavia P, Saberi S, Lakdawala NK, Wheeler MT, Owens A, Kubanek M, Wojakowski W, Jensen MK, Gimeno-Blanes J, Afshar K, Myers J, Hegde SM, Solomon SD, Sehnert AJ, Zhang D, Li W, Bhattacharya M, Edelberg JM, Waldman CB, Lester SJ, Wang A, Ho CY, Jacoby D; EXPLORER-HCM study investigators. Mavacamten for treatment of symptomatic obstructive hypertrophic cardiomyopathy (EXPLORER-HCM): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2020 Sep 12;396(10253):759-769. doi: 10.1016/S0140-6736(20)31792-X. Epub 2020 Aug 29. PMID 32871100